CLINICAL TRIAL: NCT05695339
Title: Phase I Open Label Clinical Trial Using Resiniferatoxin, A Non-Opioid Medication, For the Management of Refractory Morton's Neuroma Pain
Brief Title: Resiniferatoxin for the Management of Refractory Morton s Neuroma Pain
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10000767; 000767-CC
Record Dates: First submitted 2023-01-21; First posted 2023-01-25 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11-19

CONDITIONS: Morton's Neuroma
Keywords: Neuropathic; Forefoot; Ultra-Sound Guided; Common Plantar Digital Nerve; Perineural Injection; Trpv1; Morton's Disease
MeSH Terms: conditions — Morton Neuroma | interventions — resiniferatoxin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Resiniferatoxin (Experimental): Resiniferatoxin
  Interventions: Drug: Resiniferatoxin

INTERVENTIONS:
Drug: Resiniferatoxin — An injection of 1-2 ml bupivacaine 0.5% will be placed around the affected branch of the neuroma (aiming at its proximal end) and dorsal adjacent tissue including the skin dorsally to the neuroma. This is to prevent pain caused by any microscopic spills of RTX during the. A second local anesthetic depot will be placed 1-2 cm proximally to the injection site around the affected branch of the plantar nerve to prevent pain caused by passive current transmission by axonal RTX excitation. Following the course of the affected nerve branch and ultra-sound visualization of the injection site, 0.5-2 ml bupivacaine 0.5% will be injected perineurally. Once the site has sufficient nerve block, the required RTX dose in a solution of 0.25 ml will be injected directly proximal to the Morton s neuroma under ultra-sound visualization.

SUMMARY:
Morton s neuroma is an irritation of the nerves that affect the feet. People with this condition may have burning or shooting pain in the balls of their feet. They may also have numbness in adjacent areas. These symptoms may become more frequent and severe over time. The pain may become permanent. Current treatments tend to be short-lived, and they do not work in all people. Better treatments are needed.

Objective:

To test a study drug, resiniferatoxin (RTX), in people with Morton s neuroma.

Eligibility:

Healthy people aged 18 and older who have Morton s neuroma and have tried other standard treatments that did not ease their pain.

Design:

Participants will be involved in the study up to 4 months.

They will be screened. They will have a physical exam with blood tests. They will have a test of their heart function. They will have X-rays of their affected feet. They will have tests to assess their pain and how their feet react to touch and changes in temperature. They will complete questionnaires about their pain.

RTX is injected into the foot at the site of the nerve pain. Participants will receive a shot to numb the area before the RTX is administered. They will be monitored in the clinic for 4 hours after they receive the RTX.

Participants will receive up to 5 follow-up phone calls per week. Each call will take 5 to 10 minutes. They will be asked about their foot pain and whether they have had any side effects from the RTX.

Participants will return to the clinic 4 weeks after the treatment. Previous tests will be repeated.

DETAILED DESCRIPTION:
Study Description:

This is an interventional protocol to determine the safety and tolerability of resiniferatoxin (RTX) for treatment of pain from Morton's neuroma with a single ultrasound-guided perineural injection of (RTX). It is hypothesized that RTX will provide a long-lasting reduction of the intensity of spontaneous and evoked pain and improve daily function without interfering with other sensory modalities or motor function. The safety and efficacy of the interventional procedure will be assessed during the trial. The 3+3 design of RTX treatment will be used to assess safety and determine the Dose Limiting Toxicity (DLT). Pre- and post-procedure pain intensity assessments, including graded interference of pain with daily function and graded descriptors of neuropathic pain, will be performed to assess efficacy. This protocol is intended to test RTX as a new method for long-term relief of refractory Morton s neuroma pain. Potentially this new treatment will reduce the need for radical procedures to treat unrelenting Morton s neuroma pain.

Objectives:

Primary Objective:

-To determine the safety and tolerability of resiniferatoxin (RTX) for treatment of pain from Morton's neuroma.

Secondary Objective:

-To determine the efficacy of RTX intervention on pain intensity, interference of pain with daily function and incidence and intensity of neuropathic qualities of pain.

Endpoints:

Primary Endpoint:

-The number of related Adverse Events (Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials) experienced between day 0 (injection day) and day 28 post-injection.

Secondary Endpoints:

* Change in average worst pain (NRS) between day 21 and day 28 compared to baseline average worst pain.
* Change in pain interference on day 28 compared to screening (preinjection) using PROMIS pain tools.

Change in neuropathic pain score on day 28 compared to screening (preinjection)using painDETECT.

ELIGIBILITY:
* INCLUSION CRITERIA:

Both male and female participants are eligible for study evaluation. There are no exclusions for any racial/ethnic groups. Efforts will be made to extend accrual to a representative population. In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Provision of signed and dated informed consent form.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Must be able to read, write, understand, and complete English-language study-related forms and adequately communicate in English.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female, aged 18 and older.
* In good general health as evidenced by medical history.
* Diagnosed with one painful Morton s neuroma in the index foot
* Has not attained satisfactory pain relief with conservative, oral analgesic and at least one kind of injection treatment for Morton s neuroma.
* Exhibits moderate to severe foot pain due to the Morton s neuroma (average worst pain >= 5 on the 0-10 numeric pain rating scale NRS) as assessed verbally at >= 3 individual days during prescreening.
* For females of reproductive potential who are sexually active: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional one (1) month after administration of RTX.

If a female, be sterile (surgically or biologically) * or at least one year postmenopausal**, or have a monogamous partner who is surgically sterile, or have a same sex partner, or if in a heterosexual relationship, must agree to do the following for at least one month after receiving investigational product (IP):

* Practice abstinence, or
* Use at least one of the following medically acceptable methods of birth control:

  * Hormonal methods such as oral, implantable, injectable, vaginal ring, or transdermal contraceptives (must have started a minimum of 1 full cycle, based on the subject s usual menstrual cycle period, before IP dose
  * Intrauterine device
  * Double-barrier method (condoms, sponge, or diaphragm with spermicidal jellies or cream).

    * Defined as having had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy or bilateral tubal ligation/occlusion at least 6 weeks prior to screening; or having a congenital or acquired condition that prevents childbearing

      * Defined as at least 12 months with no menses without an alternative medical cause) [can be confirmed with follicle stimulating hormone level (FSH) in the post-menopausal range (FSH levels >=40 milli international units/mL (mIU/mL) at Screening) if the subject is not on hormonal replacement therapy]
* For males of reproductive potential who are sexually active: use of condoms or other methods to ensure effective contraception with partner for one (1) month after administration of (RTX).

If a male of reproductive potential, unless he has a same sex partner or a partner who is sterile or at least one year post-menopausal, must agree to do the following for at least one month after receiving IP

* practice abstinence from heterosexual activity or
* use (or have their partner use) acceptable contraception (see criterion above) during heterosexual activity

Male study participants should not donate sperm for 3 months after RTX injection.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Pregnancy or lactation.
* Has a known allergy or hypersensitivity to chili peppers or capsaicin.
* Has a known allergy to local anesthetics.
* Has active or history of rheumatoid arthritis or peripheral neuropathy.
* Has a prolonged baseline QTc interval exceeding 480 milliseconds.
* Current presentation of other currently painful pathology of the same foot affected by Morton s neuroma, including, but not limited to, hallux valgus, plantar fasciitis, hammer toes, metatarsalgia, bursitis.
* History of injection and/or ablation treatments treatment in the affected foot up to one month previous to study participation.
* History of nerve excision due to Morton s neuroma in the location to be treated with RTX.
* Active cutaneous disease, inflammation or infection at the anticipated site of study drug injection.
* Has diabetes mellitus or peripheral vascular disease whether poorly managed or stable.
* Has more than one Morton s neuroma in the index foot scheduled to receive the treatment intervention.
* Other clinically significant condition that might interfere with study participation or greatly increases safety risk to the subject, as judged by the study investigator.
* Concurrent treatment with another investigational drug or other intervention within last month.
* Cognitive or language difficulties that would impair comprehension or completion of the assessment instruments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The number of related Adverse Events | day 0 (injection day) and day 28 post-injection (end-of-study)
  -The number of related Adverse Events (Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials) experienced between day 0 (injection day) and day 28 post-injection
DLT or the highest dose | day 0 (injection day) and day 28 post-injection (end-of-study).
  -The number of related Adverse Events (Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials) experienced between day 0 (injection day) and day 28 post-injection

SECONDARY OUTCOMES:
Change in average worst pain (NRS) | between day 21 and 28
  Change in average worst pain (NRS) between day 21 and 28 compared to baseline average worst pain (NRS)
Change in pain interference | Day 28
  Change in pain interference on day 28 compared to screening (pre-injection) using BPI-SF
Change in neuropathic pain score | Day 28
  Change in neuropathic pain score on day 28 compared to screening (pre-injection) using painDETECT

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Mannes, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000767-CC.html